CLINICAL TRIAL: NCT03623789
Title: Blood-saving Effect of Combined Intravenous Tranexamic Acid With Topical Floseal® Application, a Comparison With Intravenous Tranexamic Acid Only in Total Hip Arthroplasty
Brief Title: Blood-saving Effect of Combined Intravenous Tranexamic Acid With Topical Floseal® Application Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201701718A3
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hip Replacement, Total
Keywords: Total hip arthroplasty; Tranexamic acid; Floseal; postoperative blood loss; Thrombin
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranylcypromine; FloSeal Matrix; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Primary total hip replacement with application of Floseal hemostatic matrix on potential bleeding sites after prosthesis implantation, and intravenous application of tranexamic acid1 g TXA before incision, followed by two boluses (1g TXA) three hours later and six hours later
  Interventions: Drug: intravenous application of tranexamic acid; Drug: Floseal hemostatic matrix
- Group II (Active Comparator): Primary total hip replacement with intravenous application of tranexamic acid1 g TXA before incision, followed by two boluses (1g TXA) three hours later and six hours later
  Interventions: Drug: intravenous application of tranexamic acid
- Group III (Placebo Comparator): Control group, neither TXA nor Floseal® will be used. Equivalent volume of normal saline injection pre- and post-operatively
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: intravenous application of tranexamic acid — intravenous application of tranexamic acid1 g TXA before incision, followed by two boluses (1g TXA) three hours later and six hours later.
  Other Names: transamine
  Arms: Group I; Group II
Drug: Floseal hemostatic matrix — application of Floseal® on potential bleeding sites after prosthesis implantation
  Other Names: Floseal
  Arms: Group I
Drug: Normal saline — Equivalent volume of saline injection before incision, followed by two boluses (1g TXA) three hours later and six hours later.
  Other Names: saline
  Arms: Group III

SUMMARY:
Total hip arthroplasty (THA) is an excellent surgical procedure for patients with end-stage hip diseases. However, THA is associated with considerable blood loss and increasing needs for allogenic blood transfusion. Tranexamic acid (TXA) was reportedly effective reducing total blood loss (TBL) after standard THA. However, a TBL of one L is still high for elderly patients.

Floseal (Baxter, Deerfield, Illinois), a thrombin-based hemostatic agent, have been widely used in surgical procedure. However, there is no study investigating the effect of Floseal in THA procedures.This study anticipated that combination with the two different mechanism of topical hemostatic agent, Floseal, and intravenous TXA can bring a synergistic blood saving effect in THA patients.

Purpose:

Our purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of combination of intravenous TXA and topical Floseal in a primary THA procedure.

Material and Methods:

The patients who are enrolled in this study will be assigned into three groups. The first group will be treated by combination of 1 g of TXA pre-operatively and two boluses TXA post-operatively intravenously and Floseal topical application, the second group by 1 g of TXA pre-operatively and two boluses TXA postoperatively intravenously without Floseal use, and the third group was control group which will be treated without TXA and Floseal. This study will observe whether there is difference in the blood-conservation effect by total blood loss calculation, hemoglobin loss and transfusion requirement between these three groups.

This study anticipate that combined use of intravenous TXA and Floseal in THA procedure is more effective in decreasing blood loss and blood transfusion than intravenous TXA application alone, and this formula do not increase the risk of thromboembolic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with osteoarthritis of the hip secondary to degeneration, inflammatory arthritis, gouty arthritis, acetabular dysplasia or osteonecrosis of the femoral head, and undergoing primary unilateral minimally invasive THA
2. Age > 18 years and < 90 years
3. Failure of medical treatment or rehabilitation.
4. Hemoglobin > 11g/dl,
5. No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

1. Preoperative Hemoglobin ≦11 g/dl
2. History of infection or intraarticular fracture of the affective hip
3. Renal function deficiency (GFR <30 ml/min/1.73m2)
4. Elevated liver enzyme (aspartate transaminase (AST)/ alanine transaminase(ALT) level are more than twice normal range) , history of liver cirrhosis, impaired liver function(elevated total bilirubin level) and coagulopathy (including long-term use anticoagulant)
5. History of deep vein thrombosis, ischemic heart disease or stroke
6. Contraindications of tranexamic acid, floseal, or rivaroxaban
7. Allergy to tranexamic acid, floseal, rivaroxaban, or the excipients
8. History of heparin-induced thrombocytopenia (HIT)
9. Coagulopathy or bleeding tendency caused by organ dysfunction, such as cirrhosis, bone marrow suppression etc.
10. Patient who have active bleeding disorder, such as intracranial hemorrhage, upper gastrointestinal bleeding, hematuria.
11. Patients with known allergies to materials of bovine origin.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Total Blood Loss | Post op day 4
  The total blood loss was calculated according to Nadler et al, which uses maximum postoperative decrease of the Hb level adjusted for weight and height of the patient. Total blood loss consists of amount of blood loss calculated from the maximum Hb loss and amount of blood transfused
Acute intraoperative Blood Loss | At the end of operation
  The intra-operative blood loss was recorded according to the volume of contents of the suction bottle and the estimated blood loss through weighing the swabs. The blood loss volume (ml) will be the volume of contents of the suction plus the increasing weight (gm) of swabs (supposing the proportion of blood is 1 gm/mL)
The change of Hemoglobin level | Preoperative day 1 to Post op day 4
  Check postoperative Hemoglobin level on postoperative day 1,2,4

SECONDARY OUTCOMES:
Blood transfusion rate | Within 3 months after operation
  We will record the event of blood transfusion, and calculate the incidence of transfusion
Thrombosis risk evaluation | Within 3 months after operation
  Detect the presence of deep-vein thrombosis of both lower limbs by duplex ultrasound study before discharge
Incidence of wound complications | Within 3 months after operation
  Wound complications including hematoma, skin necrosis and infection

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Callaghan JJ, O'Rourke MR, Liu SS. Blood management: issues and options. J Arthroplasty. 2005 Jun;20(4 Suppl 2):51-4. doi: 10.1016/j.arth.2005.03.018. PMID 15991130
- [Background] Kubota R, Nozawa M, Matsuda K, Maezawa K, Kim SG, Maeda K, Ikegami T, Hayashi K, Nagayama M, Kaneko H. Combined preoperative autologous blood donation and intra-operative cell salvage for hip surgery. J Orthop Surg (Hong Kong). 2009 Dec;17(3):288-90. doi: 10.1177/230949900901700308. PMID 20065365
- [Background] Smith LK, Williams DH, Langkamer VG. Post-operative blood salvage with autologous retransfusion in primary total hip replacement. J Bone Joint Surg Br. 2007 Aug;89(8):1092-7. doi: 10.1302/0301-620X.89B8.18736. PMID 17785752
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Newman ET, Watters TS, Lewis JS, Jennings JM, Wellman SS, Attarian DE, Grant SA, Green CL, Vail TP, Bolognesi MP. Impact of perioperative allogeneic and autologous blood transfusion on acute wound infection following total knee and total hip arthroplasty. J Bone Joint Surg Am. 2014 Feb 19;96(4):279-84. doi: 10.2106/JBJS.L.01041. PMID 24553883
- [Background] Vamvakas EC, Blajchman MA. Transfusion-related mortality: the ongoing risks of allogeneic blood transfusion and the available strategies for their prevention. Blood. 2009 Apr 9;113(15):3406-17. doi: 10.1182/blood-2008-10-167643. Epub 2009 Feb 2. PMID 19188662
- [Background] Allain JP, Stramer SL, Carneiro-Proietti AB, Martins ML, Lopes da Silva SN, Ribeiro M, Proietti FA, Reesink HW. Transfusion-transmitted infectious diseases. Biologicals. 2009 Apr;37(2):71-7. doi: 10.1016/j.biologicals.2009.01.002. Epub 2009 Feb 20. PMID 19231236
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Kazemi SM, Mosaffa F, Eajazi A, Kaffashi M, Daftari Besheli L, Bigdeli MR, Zanganeh RF. The effect of tranexamic acid on reducing blood loss in cementless total hip arthroplasty under epidural anesthesia. Orthopedics. 2010 Jan;33(1):17. doi: 10.3928/01477447-20091124-30. PMID 20055345
- [Background] McConnell JS, Shewale S, Munro NA, Shah K, Deakin AH, Kinninmonth AW. Reduction of blood loss in primary hip arthroplasty with tranexamic acid or fibrin spray. Acta Orthop. 2011 Dec;82(6):660-3. doi: 10.3109/17453674.2011.623568. Epub 2011 Oct 17. PMID 21999623
- [Background] Yue C, Kang P, Yang P, Xie J, Pei F. Topical application of tranexamic acid in primary total hip arthroplasty: a randomized double-blind controlled trial. J Arthroplasty. 2014 Dec;29(12):2452-6. doi: 10.1016/j.arth.2014.03.032. Epub 2014 Mar 29. PMID 24793893
- [Background] Chen S, Wu K, Kong G, Feng W, Deng Z, Wang H. The efficacy of topical tranexamic acid in total hip arthroplasty: a meta-analysis. BMC Musculoskelet Disord. 2016 Feb 16;17:81. doi: 10.1186/s12891-016-0923-0. PMID 26878845
- [Background] Hsu CH, Lin PC, Kuo FC, Wang JW. A regime of two intravenous injections of tranexamic acid reduces blood loss in minimally invasive total hip arthroplasty: a prospective randomised double-blind study. Bone Joint J. 2015 Jul;97-B(7):905-10. doi: 10.1302/0301-620X.97B7.35029. PMID 26130344
- [Background] Xie J, Ma J, Yao H, Yue C, Pei F. Multiple Boluses of Intravenous Tranexamic Acid to Reduce Hidden Blood Loss After Primary Total Knee Arthroplasty Without Tourniquet: A Randomized Clinical Trial. J Arthroplasty. 2016 Nov;31(11):2458-2464. doi: 10.1016/j.arth.2016.04.034. Epub 2016 May 6. PMID 27262419
- [Background] Seyednejad H, Imani M, Jamieson T, Seifalian AM. Topical haemostatic agents. Br J Surg. 2008 Oct;95(10):1197-225. doi: 10.1002/bjs.6357. PMID 18763249
- [Background] Oz MC, Rondinone JF, Shargill NS. FloSeal Matrix: new generation topical hemostatic sealant. J Card Surg. 2003 Nov-Dec;18(6):486-93. doi: 10.1046/j.0886-0440.2003.00302.x. No abstract available. PMID 14992097
- [Background] Gazzeri R, Galarza M, Alfier A. Safety biocompatibility of gelatin hemostatic matrix (Floseal and Surgiflo) in neurosurgical procedures. Surg Technol Int. 2012 Dec;22:49-54. PMID 22915500
- [Background] Clapp M, Huang JC. Use of FloSeal Sealant in the Surgical Management of Tubal Ectopic Pregnancy. Case Rep Obstet Gynecol. 2013;2013:906825. doi: 10.1155/2013/906825. Epub 2013 May 29. PMID 23819082
- [Background] Testini M, Marzaioli R, Lissidini G, Lippolis A, Logoluso F, Gurrado A, Lardo D, Poli E, Piccinni G. The effectiveness of FloSeal matrix hemostatic agent in thyroid surgery: a prospective, randomized, control study. Langenbecks Arch Surg. 2009 Sep;394(5):837-42. doi: 10.1007/s00423-009-0497-5. Epub 2009 May 7. PMID 19421770
- [Background] Di Francesco A, Flamini S, Fiori F, Mastri F. Hemostatic matrix effects on blood loss after total knee arthroplasty: A randomized controlled trial. Indian J Orthop. 2013 Sep;47(5):474-81. doi: 10.4103/0019-5413.118203. PMID 24133307
- [Background] Suarez JC, Slotkin EM, Alvarez AM, Szubski CR, Barsoum WK, Patel PD. Prospective, randomized trial to evaluate efficacy of a thrombin-based hemostatic agent in total knee arthroplasty. J Arthroplasty. 2014 Oct;29(10):1950-5. doi: 10.1016/j.arth.2014.05.025. Epub 2014 Jun 5. PMID 25015756
- [Background] Kim HJ, Fraser MR, Kahn B, Lyman S, Figgie MP. The efficacy of a thrombin-based hemostatic agent in unilateral total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2012 Jul 3;94(13):1160-5. doi: 10.2106/JBJS.K.00531. PMID 22623075
- [Background] Helito CP, Gobbi RG, Castrillon LM, Hinkel BB, Pecora JR, Camanho GL. Comparison of Floseal(r) and electrocautery in hemostasis after total knee arthroplasty. Acta Ortop Bras. 2013;21(6):320-2. doi: 10.1590/S1413-78522013000600004. PMID 24453689
- [Background] Comadoll JL, Comadoll S, Hutchcraft A, Krishnan S, Farrell K, Kreuwel HT, Bechter M. Comparison of hemostatic matrix and standard hemostasis in patients undergoing primary TKA. Orthopedics. 2012 Jun;35(6):e785-93. doi: 10.3928/01477447-20120525-14. PMID 22691647
- [Background] Bae KC, Cho CH, Lee KJ, Son ES, Lee SW, Lee SJ, Lim KH. Efficacy of intra-articular injection of thrombin-based hemostatic agent in the control of bleeding after primary total knee arthroplasty. Knee Surg Relat Res. 2014 Dec;26(4):236-40. doi: 10.5792/ksrr.2014.26.4.236. Epub 2014 Dec 2. PMID 25505706